CLINICAL TRIAL: NCT06171672
Title: The Lived Experience of Pediatric Nurse-caregiver Relationship in the PICU: a Descriptive Phenomenological Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Other Study IDs: Lived experience_PICU
Record Dates: First submitted 2023-11-20; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Intensive Care Units, Pediatric
Keywords: Nurse experience; PICU; Semi structured interview

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- semi-structured interview for nurses: Pediatric intensive care nurses in Hong Kong will be invited to join an individual in-depth semi structured interview.
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — Pediatric intensive care nurses in Hong Kong will be invited to join an individual in-depth semi structured interview.

SUMMARY:
The goal of this qualitative study is to make exploration in the lived experience of pediatric nurse-caregiver relationship in the PICU. The main question it aims to answer is:

• What is the meaning of nurse-caregiver relationship among pediatric intensive care nurses in Hong Kong

Participants will be invited to undergo individual, in-depth, semi-structured interviews.

DETAILED DESCRIPTION:
Pediatric intensive care nurses care not only for critically ill children but also for their caregivers. Under unfamiliar and critical situations, caregivers demand nursing care to ease their negative emotions and to cope. Pediatric intensive care nurse is the bridge to connect the healthcare team to the caregivers in the pediatric intensive care units (PICU). Previous literature discussed the relationship between nurses and family caregivers as therapeutic and meaningful, which consisted of elements like mutual respect, empathy, support, and more. Nurses' and family caregivers' roles shifted and changed in different times and settings. However, the relationship between the two had not been acknowledged in the PICU context. A review of the literature showed that the interaction between the pediatric intensive care nurse and the family caregivers involved six elements. Consequently, a conceptual framework was developed which may help represent the essence of the nurse-caregiver relationship.

This study aims to explore the lived experience as to the meaning of nurse-caregiver relationship among pediatric intensive care nurses in Hong Kong. Descriptive phenomenological approach will be adopted to gain an accurate and unbiased description of the lived experience. An estimated ten pediatric intensive care nurses in Hong Kong will be invited to undergo individual, in-depth, semi-structured interviews. Hence to obtain pediatric intensive care nurses' detailed information so as to reveal the essence of Nurse-Caregiver Relationship in PICU.

Data will be analyzed using Colaizzi's seven-step strategy as it aligns with the study aim and is able to obtain the meaning of experience. This qualitative study may disclose the nurse-caregiver relationship and the complex nursing relationship role in the context of PICU in Hong Kong and allow clinical reasoning to improve FCC via understanding pediatric intensive care nurses' experience.

ELIGIBILITY:
Inclusion Criteria:

* any full-time registered nurse in any hospital in Hong Kong
* interacted with the caregivers of NICU/PICU patients in the last 12 months
* with at least 12 months' experience in NICU/PICU
* able to speak in Cantonese and read Chinese
* being willing to articulate their feelings and experiences

Exclusion Criteria:

* Part-time registered nurses
* student nurses
* enrolled nurses

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Full-time registered nurse who has worked in Hong Kong with experience interating with caregives in NICU/PICU will be recruited.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interview | Data collection and analysis will be done simultaneously at day 1
  the interview will be transcribed in Cantonese after each interview

CONTACTS AND LOCATIONS:
Locations (1):
- Katherine Lam, Hong Kong, Hong Kong,China, Hong Kong